CLINICAL TRIAL: NCT00162695
Title: Rhabdomyosarcoma and Malignant Soft Tissue Tumours of Childhood
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMS95
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2005-09-13 (Estimated); Status verified 2005-09

CONDITIONS: Rhabdomyosarcoma; Malignant Soft Tissue
MeSH Terms: conditions — Rhabdomyosarcoma | interventions — Ifosfamide; Vincristine; Epirubicin; Carboplatin; Etoposide

INTERVENTIONS:
Drug: Ifosfamide, oncovin, actinomycine D, epirubicine, carboplatinum, etoposide

SUMMARY:
Objective of the study objectives was to explore survival advantage for an intensified chemotherapy strategy in a randomised trial.

IVA (ifosfamide, vincristine, actinomycin D) or a 6 drug combination (IVA + carboplatin, epirubicin, etoposide) both delivered over 27 weeks. Cumulative dose / m2 = ifosfamide 54g (both arms), epirubicin 450 mg, etoposide 1350 mg (6 drug). Delivery of radiotherapy was determined according to site and / or response to chemotherapy ± surgery.

The study was powered to detect 10% difference in 3 year OS.

ELIGIBILITY:
Inclusion Criteria:

* age > 6 months and < 18 years
* no distant metastases
* diagnosis within previous 8 weeks without prior treatment except surgery
* pathology available for central review
* written consent according to institutional requirement

Exclusion Criteria:

* stage III (node positive)
* stage I or II non alveolar orbital tumours
* patients with parameningeal disease aged < 3 years

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400
Dates: Start 1995-07

PRIMARY OUTCOMES:
To explore survival advantage for an intensified chemotherapy strategy in a randomised trial

CONTACTS AND LOCATIONS:
Overall Officials: Odile OBERLIN, Dr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Michael STEVENS, Dr, Principal Investigator — Hospital of Bristols, UK
Locations (1):
- Institut Gustave Roussy, Villejuif, France